CLINICAL TRIAL: NCT04946149
Title: Psychosocial Factors, Lifestyle and Central Pain Processing as Potential Predictors of Outcome After Rehabilitation for Rotator Cuff Repair: A Study Design for a Prospective Longitudinal Cohort Study
Brief Title: Psychosocial Factors, Lifestyle and Central Pain Processing as Potential Predictors of Outcome for Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ariane Schwank, Clinical Specialist upper extremity, Physiotherapy / Physical Therapist, Master of Science, Kantonsspital Winterthur KSW
Other Study IDs: ID2018-02089
Record Dates: First submitted 2021-06-10; First posted 2021-06-30 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Rotator Cuff Tear or Rupture, Not Specified as Traumatic
Keywords: rotator cuff repair; pain catastrophising; distress; psychological factors; expectations; sleep; central pain prossecing
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The influence of modifiable psychosocial and lifestyle factors and the role of central pain processing (CPP) on outcome after rotator cuff repair (RCR) is not well enough established to formulate holistic prognosis. Modern pain neuroscience emphasises to explain musculoskeletal shoulder pain biopsychosocially, which seems short when looking at the yearly RCR increase. This study will explore modifiable psychosocial and lifestyle factors and CPP as potential predictors for outcome after RCR.

DETAILED DESCRIPTION:
Shoulder pain is the third most common musculoskeletal disorder seen in primary care with low recovery rates (50-60%) 12 to 18 months post onset. Rotator cuff (RC) disorders are the most common amongst shoulder pain patients with a life-time prevalence of around 70%. There is a lack of consensus concerning the cause of shoulder pain, as many people present with structural changes of their RC, yet they do not suffer pain. Reports from the United States acknowledge that only one third of RC lesions are symptomatic. RC degeneration measured in cadavers, increases rapidly from the age of 50 to 55, peaking at 80 years. Contrary to this observed increasing mechanistic change, the pain curve from the age of 65 onwards. This decrease in pain implies that shoulder pain is not solely based upon the presence of a RC tear, or other underlying structural changes.

Patients who demonstrate structural changes of their RC, are still predominantly treated using biomedical reasoning. There was a reported 270,000 annual surgeries in the USA and an increase of 204% in rotator cuff repairs (RCR) between 1998 and 2011 in Finland. Satisfactory outcomes ranged from 38% to 95%. Biomedical prognostic indicators dominate the orthopaedic research on outcomes post RCR. Biomedical factors include; arm function (e.g. muscle strength), radiological findings (e.g. tear size) or demographics (e.g. age). This assertion was backed by a systematic review and meta-analysis regarding prognosis post RCR, where mainly anatomical and functional shoulder factors were analysed.

Despite the reliance on biomedical indicators, there is a growing body of evidence about the impact of psychosocial factors on persistent shoulder pain, and on outcomes after RCR. The biopsychosocial model first described by Engel in the 1970's incorporates multiple dimensions and explains illness or disease based upon biomedical, psychological and social determinants of health. The perception of high job demand, poor social support, baseline high distress, maladaptive pain beliefs such as catastrophic thinking and pain self-efficacy can lead to persistent shoulder pain and disability. The absence of psychological distress is also associated with improved self-efficacy ("the capacity to produce important effects"), and lower levels of pain and disability. However, studies on the influence of psychosocial factors post RCR, demonstrate weak interactions. Patients with existing preoperative psychological conditions like depression and anxiety or cognitive psychological factors like pain catastrophizing and kinesiophobia, and psychological distress demonstrate higher pre-operative pain levels.

High patients' expectations of a positive outcome post RCR show independent and strong associations to satisfactory outcomes after RCR, measured in pain and disability, and performance at one-year post-op. However, it is unclear which circumstances lead to high or low expectations and how one should measure these. Low expectations in conservative treatments like physiotherapy, can be influenced by the patients' biomedical oriented attitudes and beliefs towards pain and disability. High expectations on outcome post RCR may be further driven by the failure of conservative treatments (e.g. Physiotherapy).

Sleep disturbance is highly prevalent in rotator cuff related shoulder pain patients and shoulder pain was found to be a strong predictor for sleep disturbance. RCR seems to reduce this vicious interplay between pain and sleep as findings demonstrate an overall post RCR improvement of sleep quality. The same study did not find any predictive power for insomnia on outcome post RCR.

The relationship between CPP measures such as central sensitisation (CS), or quantitative sensory testing (QST) and prolonged shoulder pain have been established.

To conclude, in the literature there is a lack of knowledge about modifiable psychosocial and lifestyle factors and CPP for predicting outcome after RCR. Clinicians need an improved explanatory model to predict successful outcomes post RCR. Neither the local tissue pathology-pain model nor the growing knowledge about local biochemical changes in the tendons, sufficiently describe the relationship between tissue changes and perceived shoulder pain. There is insufficient understanding to what extent cognitive psychological factors like pain catastrophizing, high perceived stress or low self-efficacy may influence outcome after RCR and whether or not they drive high or low patients' expectations (psychosocial factor) for surgery. The role of sleep on outcome after RCR remains obscure. Finally, the association of CPP with prolonged recovery post RCR is unknown.

This study aims to support the understanding of psychosocial factors and their influence on outcome after RCR. The investigators hypothesise that psychosocial factors, lifestyle factors and CPP do play a role in individual prognosis for outcome after RCR. If modifiable psychosocial or lifestyle related factors such as patients' expectations on surgery, catastrophic pain thinking, high perceived stress, altered injury perceptions, sleep disturbance or altered central pain processing are identified as predictors for post RCR outcome, clinicians might tailor treatment and potentially patient selection for RCR based upon improved factors and hypothetically reduce the number of persistent shoulder pain patients one year after onset.

This study aims to answer the following questions:

1. Is there an association between psychosocial factors including expectations, lifestyle factors such as sleep and CPP with outcome (quality of life, pain and disability) after RCR at 12 weeks and 12 months?
2. To what extent do these pre-interventional variables predict post-operative RCR outcome at 12 weeks and 12 months? Methods Study Design and setting The study will be implemented and reported in line with the STROBE statement for observational studies.

Data are obtained monocentric in the shoulder and elbow surgery unit in the clinic of orthopaedic surgery and traumatology in alliance with the institute of therapy and rehabilitation of the acute care hospital, "Kantonsspital Winterthur" in Switzerland.

The current research project will analyze data from three selected time points of this clinical routine of the RCR management; 2-3 weeks preoperative (T1), 12 weeks postoperative (T2) and 12 months postoperative (T3). Data from January 2019 will be considered. Data collection will be stopped after the inclusion of 141 individual datasets with 12 months follow up, estimated to be completed in late Spring 2022.

Demographic variables such as age, gender, and profession and comorbidities, including diabetes, rheumatological disease, cardiovascular disease, and neurological disease, will be registered.

The investigators will use a mixed-effects regression model for repeated measures. This will have the power to detect a moderate effect size that is still clinically relevant (15% difference in WORC score) with confidence level α=0.5, (two-tailed) and a desired power of 90%. The required total sample size was calculated to be 125 subjects (Edland). Mixed models do not require complete datasets to produce accurate results, but the statistical analysts have accounted for potential attrition. Given an expected drop-out rate of approximately 12.5%, a total number of 141 patients is needed. The power is set at 90% to minimize the chance of making a type II error.

Statistical Methods and Analysis Statistical analyses will be performed using RStudio. Level of significance is set at p = 0.05. Appropriate descriptive statistics will be performed. Measurements will take place at three time points in the perioperative management, as described above (T1 = at baseline 2-3 weeks prior to RCR, T2 = at 12 weeks post RCR and T3 = at 12 months post RCR as follow-up).

The primary outcome (WORC) will be analysed using multilevel linear regression models for repeated (longitudinal) measures, using an unstructured covariance matrix. Dependent variables are the primary and secondary outcomes. Continuous secondary outcomes will be assessed in a similar way to the primary outcome. The models will be developed by stepwise reduction of the potential predictors (for, psychosocial factors, sleep and CPP). Categorical data (e.g. EQ-5D-5L) will be analysed using logistic models. For non-repeated continuous and binary measurements, ordinary linear regression and logistic models will be used, respectively. Six predictors as clustered variables will be studied. The psychosocial variables are: 1) expectation, 2) pain catastrophizing, 3) perceived stress, 4) illness perceptions; the lifestyle factor; 5) sleep and 6) central pain processing (see table 2 for more detail).

Data security and management Data generation, transmission, storage and analysis within this project strictly follow Swiss legal requirements for data protection. The electronic data capture (EDC) software REDCap (www.project---redcap.org) will be used for data processing and management. Appropriate coded identification (e.g. pseudonymisation) is used in order to enter subject data into the database. The coding list of target data is saved in a secured folder on the hospital's server.

Ethics The study underlies the principles of the Helsinki Declaration. Only data of patients who gave general consent to the hospital or informed written consent to the project will be considered for analysis. Ethical approval received January 2019 (ID 2018-02089) by the Ethical Committee of the Canton of Zurich, Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective arthroscopic RCR;
* First time RCR on the target shoulder;
* Completed primary and secondary outcome measures (Western Ontario Rotator Cuff Index (WORC), Constant Score, Maximum Pain on Numeric Rating Scale and EQ-5D-5L) from daily routine.

Exclusion Criteria:

* Changes of intra operative procedure (e.g. anything but RCR)
* Re-repair of tendon;
* No surgery;
* Other pain-related or neurological comorbidities that could interfere with pain measures;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult musculoskelettal shoulder pain patients, scheduled for first time rotator cuff repair at the acute care hospital Kantonsspital Winterthur in Switzerland.
  Traumatic and non-traumatic origin of shoulder pain.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) change from preOP to 12 weeks postOP and preOP to 12months postOP | pre operative (T1), 12 Weeks postoperative (T2), 12 months postoperative (T3)
  This 21 - items self-reported questionnaire represents a quality of life measure in rotator cuff pathology. The WORC measures 5 dimensions (pain, sports/leisure, work, daily living, feelings) with 3-6 questions per domain, measured on a 100mm Visual Analogue Scale (VAS). Left endpoint equals "no" and right endpoint equals "extreme". The total WORC score ranges from 0 (best) to 2100 (worst) (21 items x 100mm). The minimal important difference (MID) is calculated at 300mm. The PROM is reported to have positive evidence for 5 psychometric properties; internal consistency, reliability, content validity, hypothesis testing and responsiveness.

SECONDARY OUTCOMES:
Constant-Murlex Score change from preOP to 12months postOP | pre operative (T1), 12 months postoperative (T3)
  The Constant-Murley Score assesses shoulder function of which 35 % are subjective variables (maximum pain intensity, work, sport/leisure, sleep, pain free height for light work), and 65% are objective variables (range of motion (ROM) and strength measure). A sum score of 100 represents perfect shoulder function, 0 represents no functionality
Maximum Pain on Numeric Rating Scale (NRS), change from preOP to 12 weeks postOP and preOP to 12months postOP | pre operative (T1), 12 Weeks postoperative (T2), 12 months postoperative (T3)
  Patients are asked to indicate the maximum perceived shoulder pain felt in daily life on an NRS from 0 (no pain at all) to 10 (worst imaginable pain)
EQ-5D-5L, Euroqol 5dimensions, 5 levels, Quality of life measure, change from preOP to 12 weeks postOP and preOP to 12months postOP | pre operative (T1), 12 Weeks postoperative (T2), 12 months postoperative (T3)
  The research group EuroQol developed the EQ-5D-5L tool "in order to provide a simple, generic measure of health for clinical and economic appraisal". It contains of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and depression/anxiety and 5 levels ranging from no problems, slight problems, moderate problems, severe problems, and extreme problems.
Subjective Shoulder Value, change from preOP to 12 weeks postOP and preOP to 12months postOP | pre operative (T1), 12 Weeks postoperative (T2),12 months postoperative (T3)
  The SSV is evaluated by one single standardised question:" What is the overall percent value of your shoulder, if a completely normal shoulder represents 100%?"

OTHER OUTCOMES:
Potential predictor: Central pain processing: Central sensitization inventory | pre operative (T1)
  The original English questionnaire was developed in 2011 to assess key symptoms in relation to central sensitivity symptoms (CSS). It consists of two parts; Part A with 25 items relating to pain, psychosocial aspects, cognitive and functional aspects. Part B with 7 different CSSs, like restless legs, irritable bowel, and multiple chemical sensitivities and 3 disorders like neck pain (whiplash), depression and anxiety or panic attacks.
  It is a high-quality measurement tool, with high construct validity and test-retest reliability. The defined cut-off point is at 40 points.
Potential predictor: Central pain processing: Central sensitization inventory | 12 Weeks postoperative (T2)
  The original English questionnaire was developed in 2011 to assess key symptoms in relation to central sensitivity symptoms (CSS). It consists of two parts; Part A with 25 items relating to pain, psychosocial aspects, cognitive and functional aspects. Part B with 7 different CSSs, like restless legs, irritable bowel, and multiple chemical sensitivities and 3 disorders like neck pain (whiplash), depression and anxiety or panic attacks.
  It is a high-quality measurement tool, with high construct validity and test-retest reliability. The defined cut-off point is at 40 points.
Potential predictor: Central pain processing: Central sensitization inventory | 12 months postoperative (T3)
  The original English questionnaire was developed in 2011 to assess key symptoms in relation to central sensitivity symptoms (CSS). It consists of two parts; Part A with 25 items relating to pain, psychosocial aspects, cognitive and functional aspects. Part B with 7 different CSSs, like restless legs, irritable bowel, and multiple chemical sensitivities and 3 disorders like neck pain (whiplash), depression and anxiety or panic attacks.
  It is a high-quality measurement tool, with high construct validity and test-retest reliability. The defined cut-off point is at 40 points.
Potential predictor: Central pain processing: Quantitative Sensory Testing: cold hyperalgesia | pre operative (T1)
  Cold hyperalgesia is measured with a cold pack. The cold application is kept for 10 seconds, and the patients will rate the experienced pain on a NRS from 0 (no pain at all) to 10 (worst imaginable pain).
Potential predictor: Central pain processing: Quantitative Sensory Testing: cold hyperalgesia | 12 Weeks postoperative (T2)
  Cold hyperalgesia is measured with a cold pack. The cold application is kept for 10 seconds, and the patients will rate the experienced pain on a NRS from 0 (no pain at all) to 10 (worst imaginable pain).
Potential predictor: Central pain processing: Quantitative Sensory Testing: cold hyperalgesia | 12 months postoperative (T3)
  Cold hyperalgesia is measured with a cold pack. The cold application is kept for 10 seconds, and the patients will rate the experienced pain on a NRS from 0 (no pain at all) to 10 (worst imaginable pain).
Potential predictor: Central pain processing: Quantitative Sensory Testing: Pressure Pain Threshold | pre operative (T1)
  Pressure Pain Threshold (PPT): The measurements will be conducted by digital hand-held pressure algometer with a rubber tip of approximately 1 cm² (FPX 50, FORCE TEN by Wagner Instruments), increasing pressure will be given perpendicular to the skin . Measurements are taken at five standardized sites. .
Potential predictor: Central pain processing: Quantitative Sensory Testing: Pressure Pain Threshold | 12 Weeks postoperative (T2)
  Pressure Pain Threshold (PPT): The measurements will be conducted by digital hand-held pressure algometer with a rubber tip of approximately 1 cm² (FPX 50, FORCE TEN by Wagner Instruments), increasing pressure will be given perpendicular to the skin . Measurements are taken at five standardized sites. .
Potential predictor: Central pain processing: Quantitative Sensory Testing: Pressure Pain Threshold | 12 months postoperative (T3)
  Pressure Pain Threshold (PPT): The measurements will be conducted by digital hand-held pressure algometer with a rubber tip of approximately 1 cm² (FPX 50, FORCE TEN by Wagner Instruments), increasing pressure will be given perpendicular to the skin . Measurements are taken at five standardized sites. .
Potential predictor: Central pain processing: Quantitative Sensory Testing: Temporal Summation | pre operative (T1)
  Measurement tool is a Frey Filament / monofilament calibrated to 10g. The patient is asked to rate the first touch on an NRS from 0 (no pain at all) to 10 (worst imaginable pain). Then the measurement is repeated once per second (1Hz) for 30seconds on a surface of maximum 1cm2. After the 30 seconds application, the patient is asked to rate the last touch on an NRS. The difference between the last and the first rating is calculated. Fifteen seconds after the test, patients need to rate any ongoing pain sensation on NRS again.
Potential predictor: Central pain processing: Quantitative Sensory Testing: Temporal Summation | 12 Weeks postoperative (T2)
  Measurement tool is a Frey Filament / monofilament calibrated to 10g. The patient is asked to rate the first touch on an NRS from 0 (no pain at all) to 10 (worst imaginable pain). Then the measurement is repeated once per second (1Hz) for 30seconds on a surface of maximum 1cm2. After the 30 seconds application, the patient is asked to rate the last touch on an NRS. The difference between the last and the first rating is calculated. Fifteen seconds after the test, patients need to rate any ongoing pain sensation on NRS again.
Potential predictor: Central pain processing: Quantitative Sensory Testing: Temporal Summation | 12 months postoperative (T3)
  Measurement tool is a Frey Filament / monofilament calibrated to 10g. The patient is asked to rate the first touch on an NRS from 0 (no pain at all) to 10 (worst imaginable pain). Then the measurement is repeated once per second (1Hz) for 30seconds on a surface of maximum 1cm2. After the 30 seconds application, the patient is asked to rate the last touch on an NRS. The difference between the last and the first rating is calculated. Fifteen seconds after the test, patients need to rate any ongoing pain sensation on NRS again.
Potential predictor: psychosocial factor: expectation | pre operative (T1)
  Patients' expectations will be assessed using 5 questions adopted from the literature studying the Musculoskeletal Outcomes Data Evaluation and Management System (MODEMS) questionnaire among others.
Potential predictor: psychosocial factor: Pain Catastrophizing scale | pre operative (T1)
  The Pain Catastrophizing Scale assesses whether or not there is presence of catastrophic thinking about pain. Thirteen items entail aspects about different thoughts and feelings whilst experiencing pain. Items are scored on a 5-point Likert scale. Higher scores indicate more severe catastrophic thinking about pain. There is a total score and a score for three subscales (e.g. helplessness, magnification and rumination). The included German version showed similar psychometric properties like the original English version.
Potential predictor: psychosocial factor: Pain Catastrophizing scale | 12 Weeks postoperative (T2)
  The Pain Catastrophizing Scale assesses whether or not there is presence of catastrophic thinking about pain. Thirteen items entail aspects about different thoughts and feelings whilst experiencing pain. Items are scored on a 5-point Likert scale. Higher scores indicate more severe catastrophic thinking about pain. There is a total score and a score for three subscales (e.g. helplessness, magnification and rumination). The included German version showed similar psychometric properties like the original English version.
Potential predictor: psychosocial factor: Pain Catastrophizing scale | 12 months postoperative (T3)
  The Pain Catastrophizing Scale assesses whether or not there is presence of catastrophic thinking about pain. Thirteen items entail aspects about different thoughts and feelings whilst experiencing pain. Items are scored on a 5-point Likert scale. Higher scores indicate more severe catastrophic thinking about pain. There is a total score and a score for three subscales (e.g. helplessness, magnification and rumination). The included German version showed similar psychometric properties like the original English version.
Potential predictor: psychosocial factor: Perceived Stress Scale | pre operative (T1)
  The Perceived Stress Scale (PSS - 10) includes 10 questions and assesses the degree to which life has been experienced as unpredictable, uncontrollable and overloaded in the past months. The questions are answered by "yes" or "no". According to the developers of the questionnaire, perceived stress is a unidimensional construct. The questions are general in nature and therefore the usage for the cohort present in this study is reasonable. The German version showed good psychometric properties (validity and reliability)
Potential predictor: psychosocial factor: Perceived Stress Scale | 12 Weeks postoperative (T2)
  The Perceived Stress Scale (PSS - 10) includes 10 questions and assesses the degree to which life has been experienced as unpredictable, uncontrollable and overloaded in the past months. The questions are answered by "yes" or "no". According to the developers of the questionnaire, perceived stress is a unidimensional construct. The questions are general in nature and therefore the usage for the cohort present in this study is reasonable. The German version showed good psychometric properties (validity and reliability)
Potential predictor: psychosocial factor: Perceived Stress Scale | 12 months postoperative (T3)
  The Perceived Stress Scale (PSS - 10) includes 10 questions and assesses the degree to which life has been experienced as unpredictable, uncontrollable and overloaded in the past months. The questions are answered by "yes" or "no". According to the developers of the questionnaire, perceived stress is a unidimensional construct. The questions are general in nature and therefore the usage for the cohort present in this study is reasonable. The German version showed good psychometric properties (validity and reliability)
Potential predictor: psychosocial factor: Illness perception questionnaire | pre operative (T1)
  The Illness Perception Questionnaire Revised (IPQ-R) is designed to assess the cognitive and emotional representations of illness. So called illness perceptions are described as patients' cognitions about their illness, which are formed by experiences, provided information and interpretation of symptoms. The IPQ-R is not disease specific and may be used in any group of interest. It assesses 9 dimensions of illness perceptions and includes 3 domains cited by from Lau et al. (1989). The first domain is called illness identity, the second is called the beliefs domain and the third is labelled as the consequence domain. The answers are captured on a 5-point Likert scale from "strongly disagree" to "strongly agree". The clinimetric properties for musculoskeletal pain are reported to be sufficient, but the questionnaire is only tested on a few musculoskeletal disorders.
Potential predictor: psychosocial factor: Illness perception questionnaire | 12 Weeks postoperative (T2)
  The Illness Perception Questionnaire Revised (IPQ-R) is designed to assess the cognitive and emotional representations of illness. So called illness perceptions are described as patients' cognitions about their illness, which are formed by experiences, provided information and interpretation of symptoms. The IPQ-R is not disease specific and may be used in any group of interest. It assesses 9 dimensions of illness perceptions and includes 3 domains cited by from Lau et al. (1989). The first domain is called illness identity, the second is called the beliefs domain and the third is labelled as the consequence domain. The answers are captured on a 5-point Likert scale from "strongly disagree" to "strongly agree". The clinimetric properties for musculoskeletal pain are reported to be sufficient, but the questionnaire is only tested on a few musculoskeletal disorders.
Potential predictor: psychosocial factor: Illness perception questionnaire | 12 months postoperative (T3)
  The Illness Perception Questionnaire Revised (IPQ-R) is designed to assess the cognitive and emotional representations of illness. So called illness perceptions are described as patients' cognitions about their illness, which are formed by experiences, provided information and interpretation of symptoms. The IPQ-R is not disease specific and may be used in any group of interest. It assesses 9 dimensions of illness perceptions and includes 3 domains cited by from Lau et al. (1989). The first domain is called illness identity, the second is called the beliefs domain and the third is labelled as the consequence domain. The answers are captured on a 5-point Likert scale from "strongly disagree" to "strongly agree". The clinimetric properties for musculoskeletal pain are reported to be sufficient, but the questionnaire is only tested on a few musculoskeletal disorders.
Potential predictor: Sleep | pre operative (T1)
  4 Questions regarding sleep quality, sleep efficiency, sleep disturbance, number of awakenings per night. The first question is transformed from the Pittsburgh Sleep Quality Index (PSQI), for sleep quality and is rated on a 4-point Likert Scale. The question 2 to 3 are formulated by suggestion from the study by Nijs et al. and adapted to shoulder pain by the first author.
Potential predictor: Sleep | 12 Weeks postoperative (T2)
  4 Questions regarding sleep quality, sleep efficiency, sleep disturbance, number of awakenings per night. The first question is transformed from the Pittsburgh Sleep Quality Index (PSQI), for sleep quality and is rated on a 4-point Likert Scale. The question 2 to 3 are formulated by suggestion from the study by Nijs et al. and adapted to shoulder pain by the first author.
Potential predictor: Sleep | 12 months postoperative (T3)
  4 Questions regarding sleep quality, sleep efficiency, sleep disturbance, number of awakenings per night. The first question is transformed from the Pittsburgh Sleep Quality Index (PSQI), for sleep quality and is rated on a 4-point Likert Scale. The question 2 to 3 are formulated by suggestion from the study by Nijs et al. and adapted to shoulder pain by the first author.
Global Rating of Change GRoC | 12 Weeks postoperative (T2)
  GRoC represents an anchor of change, not a true change. GRoC is simple and easy to administer. It is recommended to include an 11-point scale with endpoints at -5 and +5, with -5 = "very much worse", 0 = "no change" and +5 = "completely recovered". The recommendation for the single question asked by the assessor is: "With respect to your shoulder problem, how would you describe yourself now compared to pre-surgery?"
Global Rating of Change GRoC | 12 months postoperative (T3)
  GRoC represents an anchor of change, not a true change. GRoC is simple and easy to administer. It is recommended to include an 11-point scale with endpoints at -5 and +5, with -5 = "very much worse", 0 = "no change" and +5 = "completely recovered". The recommendation for the single question asked by the assessor is: "With respect to your shoulder problem, how would you describe yourself now compared to pre-surgery?"
Postoperative satisfaction survey | 12 months postoperative (T3)
  The postoperative satisfaction survey consists different grades of satisfaction. This seems relevant for analyses of the construct. The survey has not been validated in German language and therefore had to be integrated in this study by the first authors translation.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Schwank, MSc, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Coronado RA, Seitz AL, Pelote E, Archer KR, Jain NB. Are Psychosocial Factors Associated With Patient-reported Outcome Measures in Patients With Rotator Cuff Tears? A Systematic Review. Clin Orthop Relat Res. 2018 Apr;476(4):810-829. doi: 10.1007/s11999.0000000000000087. PMID 29481342
- [Background] Vincent K, Leboeuf-Yde C, Gagey O. Are degenerative rotator cuff disorders a cause of shoulder pain? Comparison of prevalence of degenerative rotator cuff disease to prevalence of nontraumatic shoulder pain through three systematic and critical reviews. J Shoulder Elbow Surg. 2017 May;26(5):766-773. doi: 10.1016/j.jse.2016.09.060. Epub 2017 Jan 12. PMID 28089260
- [Background] Bury J, Littlewood C. Rotator cuff disorders: a survey of current (2016) UK physiotherapy practice. Shoulder Elbow. 2018 Jan;10(1):52-61. doi: 10.1177/1758573217717103. Epub 2017 Jul 11. PMID 29276538
- [Background] Jain NB, Higgins LD, Losina E, Collins J, Blazar PE, Katz JN. Epidemiology of musculoskeletal upper extremity ambulatory surgery in the United States. BMC Musculoskelet Disord. 2014 Jan 8;15:4. doi: 10.1186/1471-2474-15-4. PMID 24397703
- [Background] Paloneva J, Lepola V, Aarimaa V, Joukainen A, Ylinen J, Mattila VM. Increasing incidence of rotator cuff repairs--A nationwide registry study in Finland. BMC Musculoskelet Disord. 2015 Aug 12;16:189. doi: 10.1186/s12891-015-0639-6. PMID 26265152
- [Background] Novoa-Boldo A, Gulotta LV. Expectations Following Rotator Cuff Surgery. Curr Rev Musculoskelet Med. 2018 Mar;11(1):162-166. doi: 10.1007/s12178-018-9470-7. PMID 29435813
- [Background] Henn RF 3rd, Kang L, Tashjian RZ, Green A. Patients' preoperative expectations predict the outcome of rotator cuff repair. J Bone Joint Surg Am. 2007 Sep;89(9):1913-9. doi: 10.2106/JBJS.F.00358. PMID 17768186
- [Background] Lambers Heerspink FO, Dorrestijn O, van Raay JJ, Diercks RL. Specific patient-related prognostic factors for rotator cuff repair: a systematic review. J Shoulder Elbow Surg. 2014 Jul;23(7):1073-80. doi: 10.1016/j.jse.2014.01.001. Epub 2014 Apr 13. PMID 24725900
- [Background] Cho CH, Song KS, Hwang I, Warner JJ. Does Rotator Cuff Repair Improve Psychologic Status and Quality of Life in Patients With Rotator Cuff Tear? Clin Orthop Relat Res. 2015 Nov;473(11):3494-500. doi: 10.1007/s11999-015-4258-1. PMID 25791445
- [Background] Raman J, Walton D, MacDermid JC, Athwal GS. Predictors of outcomes after rotator cuff repair-A meta-analysis. J Hand Ther. 2017 Jul-Sep;30(3):276-292. doi: 10.1016/j.jht.2016.11.002. Epub 2017 Feb 23. PMID 28237073
- [Background] Woollard JD, Bost JE, Piva SR, Kelley Fitzgerald G, Rodosky MW, Irrgang JJ. The ability of preoperative factors to predict patient-reported disability following surgery for rotator cuff pathology. Disabil Rehabil. 2017 Oct;39(20):2087-2096. doi: 10.1080/09638288.2016.1219396. Epub 2016 Aug 22. PMID 27548366
- [Background] Thorpe AM, O'Sullivan PB, Mitchell T, Hurworth M, Spencer J, Booth G, Goebel S, Khoo P, Tay A, Smith A. Are Psychologic Factors Associated With Shoulder Scores After Rotator Cuff Surgery? Clin Orthop Relat Res. 2018 Oct;476(10):2062-2073. doi: 10.1097/CORR.0000000000000389. PMID 30179945
- [Background] Noten S, Struyf F, Lluch E, D'Hoore M, Van Looveren E, Meeus M. Central Pain Processing in Patients with Shoulder Pain: A Review of the Literature. Pain Pract. 2017 Feb;17(2):267-280. doi: 10.1111/papr.12502. Epub 2016 Oct 14. PMID 27739242
- [Background] Sanchis MN, Lluch E, Nijs J, Struyf F, Kangasperko M. The role of central sensitization in shoulder pain: A systematic literature review. Semin Arthritis Rheum. 2015 Jun;44(6):710-6. doi: 10.1016/j.semarthrit.2014.11.002. Epub 2014 Nov 13. PMID 25523242
- [Background] Martinez-Calderon J, Meeus M, Struyf F, Miguel Morales-Asencio J, Gijon-Nogueron G, Luque-Suarez A. The role of psychological factors in the perpetuation of pain intensity and disability in people with chronic shoulder pain: a systematic review. BMJ Open. 2018 Apr 13;8(4):e020703. doi: 10.1136/bmjopen-2017-020703. PMID 29654040
- [Background] Kusnanto H, Agustian D, Hilmanto D. Biopsychosocial model of illnesses in primary care: A hermeneutic literature review. J Family Med Prim Care. 2018 May-Jun;7(3):497-500. doi: 10.4103/jfmpc.jfmpc_145_17. PMID 30112296
- [Background] Potter MQ, Wylie JD, Greis PE, Burks RT, Tashjian RZ. Psychological distress negatively affects self-assessment of shoulder function in patients with rotator cuff tears. Clin Orthop Relat Res. 2014 Dec;472(12):3926-32. doi: 10.1007/s11999-014-3833-1. Epub 2014 Jul 31. PMID 25080266
- [Background] Dunn WR, Kuhn JE, Sanders R, An Q, Baumgarten KM, Bishop JY, Brophy RH, Carey JL, Harrell F, Holloway BG, Jones GL, Ma CB, Marx RG, McCarty EC, Poddar SK, Smith MV, Spencer EE, Vidal AF, Wolf BR, Wright RW; MOON Shoulder Group. 2013 Neer Award: predictors of failure of nonoperative treatment of chronic, symptomatic, full-thickness rotator cuff tears. J Shoulder Elbow Surg. 2016 Aug;25(8):1303-11. doi: 10.1016/j.jse.2016.04.030. PMID 27422460
- [Background] Lawrence C, Zmistowski BM, Lazarus M, Abboud J, Williams G, Namdari S. Expectations of Shoulder Surgery Are Not Altered by Surgeon Counseling of the Patient. Joints. 2017 Aug 11;5(3):133-137. doi: 10.1055/s-0037-1605585. eCollection 2017 Sep. PMID 29270541
- [Background] Cho CH, Jung SW, Park JY, Song KS, Yu KI. Is shoulder pain for three months or longer correlated with depression, anxiety, and sleep disturbance? J Shoulder Elbow Surg. 2013 Feb;22(2):222-8. doi: 10.1016/j.jse.2012.04.001. Epub 2012 Jun 26. PMID 22738644
- [Background] Gwilym SE, Oag HC, Tracey I, Carr AJ. Evidence that central sensitisation is present in patients with shoulder impingement syndrome and influences the outcome after surgery. J Bone Joint Surg Br. 2011 Apr;93(4):498-502. doi: 10.1302/0301-620X.93B4.25054. PMID 21464489
- [Background] Valencia C, Fillingim RB, Bishop M, Wu SS, Wright TW, Moser M, Farmer K, George SZ. Investigation of central pain processing in postoperative shoulder pain and disability. Clin J Pain. 2014 Sep;30(9):775-86. doi: 10.1097/AJP.0000000000000029. PMID 24042347
- [Background] Lewis J, O'Sullivan P. Is it time to reframe how we care for people with non-traumatic musculoskeletal pain? Br J Sports Med. 2018 Dec;52(24):1543-1544. doi: 10.1136/bjsports-2018-099198. Epub 2018 Jun 25. No abstract available. PMID 29941618
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Ann Intern Med. 2007 Oct 16;147(8):573-7. doi: 10.7326/0003-4819-147-8-200710160-00010. PMID 17938396
- [Background] Buchbinder R, Page MJ, Huang H, Verhagen AP, Beaton D, Kopkow C, Lenza M, Jain NB, Richards B, Richards P, Voshaar M, van der Windt D, Gagnier JJ; Shoulder Core Outcome Set Special Interest Group. A Preliminary Core Domain Set for Clinical Trials of Shoulder Disorders: A Report from the OMERACT 2016 Shoulder Core Outcome Set Special Interest Group. J Rheumatol. 2017 Dec;44(12):1880-1883. doi: 10.3899/jrheum.161123. Epub 2017 Jan 15. PMID 28089972
- [Background] Huber W, Hofstaetter JG, Hanslik-Schnabel B, Posch M, Wurnig C. [Translation and psychometric testing of the Western Ontario Rotator Cuff Index (WORC) for use in Germany]. Z Orthop Ihre Grenzgeb. 2005 Jul-Aug;143(4):453-60. doi: 10.1055/s-2005-836677. German. PMID 16118762
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327
- [Background] Maxwell S, Sterling M. An investigation of the use of a numeric pain rating scale with ice application to the neck to determine cold hyperalgesia. Man Ther. 2013 Apr;18(2):172-4. doi: 10.1016/j.math.2012.07.004. Epub 2012 Aug 11. PMID 22892206
- [Background] Moloney N, Hall T, Doody C. An investigation of somatosensory profiles in work related upper limb disorders: a case-control observational study protocol. BMC Musculoskelet Disord. 2010 Jan 30;11:22. doi: 10.1186/1471-2474-11-22. PMID 20113518
- [Background] Walton DM, Macdermid JC, Nielson W, Teasell RW, Reese H, Levesque L. Pressure pain threshold testing demonstrates predictive ability in people with acute whiplash. J Orthop Sports Phys Ther. 2011 Sep;41(9):658-65. doi: 10.2519/jospt.2011.3668. Epub 2011 Sep 1. PMID 21885908
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Scerbo T, Colasurdo J, Dunn S, Unger J, Nijs J, Cook C. Measurement Properties of the Central Sensitization Inventory: A Systematic Review. Pain Pract. 2018 Apr;18(4):544-554. doi: 10.1111/papr.12636. Epub 2017 Nov 20. PMID 28851012
- [Background] Timmerman H, Steegers MAH, Huygen FJPM, Goeman JJ, van Dasselaar NT, Schenkels MJ, Wilder-Smith OHG, Wolff AP, Vissers KCP. Investigating the validity of the DN4 in a consecutive population of patients with chronic pain. PLoS One. 2017 Nov 30;12(11):e0187961. doi: 10.1371/journal.pone.0187961. eCollection 2017. PMID 29190718
- [Background] Meyer K, Sprott H, Mannion AF. Cross-cultural adaptation, reliability, and validity of the German version of the Pain Catastrophizing Scale. J Psychosom Res. 2008 May;64(5):469-78. doi: 10.1016/j.jpsychores.2007.12.004. PMID 18440399
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Broadbent E, Wilkes C, Koschwanez H, Weinman J, Norton S, Petrie KJ. A systematic review and meta-analysis of the Brief Illness Perception Questionnaire. Psychol Health. 2015;30(11):1361-85. doi: 10.1080/08870446.2015.1070851. Epub 2015 Aug 26. PMID 26181764
- [Background] Leysen M, Nijs J, Meeus M, Paul van Wilgen C, Struyf F, Vermandel A, Kuppens K, Roussel NA. Clinimetric properties of illness perception questionnaire revised (IPQ-R) and brief illness perception questionnaire (Brief IPQ) in patients with musculoskeletal disorders: A systematic review. Man Ther. 2015 Feb;20(1):10-7. doi: 10.1016/j.math.2014.05.001. Epub 2014 May 14. PMID 25435470
- [Background] Collins GH, Crawford SJ. Sarcocystis in goats: prevalence and transmission. N Z Vet J. 1978 Nov;26(11):288. doi: 10.1080/00480169.1978.34571. No abstract available. PMID 109801
- [Background] Blackwell E, de Leon CF, Miller GE. Applying mixed regression models to the analysis of repeated-measures data in psychosomatic medicine. Psychosom Med. 2006 Nov-Dec;68(6):870-8. doi: 10.1097/01.psy.0000239144.91689.ca. Epub 2006 Nov 1. PMID 17079709
- [Background] Edland SD, Ard MC, Sridhar J, Cobia D, Martersteck A, Mesulam MM, Rogalski EJ. Proof of concept demonstration of optimal composite MRI endpoints for clinical trials. Alzheimers Dement (N Y). 2016 Sep;2(3):177-181. doi: 10.1016/j.trci.2016.05.002. PMID 28345017
- [Derived] Schwank A, Struyf F, Struyf T, Mertens M, Gisi D, Benninger E, Meeus M. Psychosocial Factors, Sleep, and Central Pain Processing for Making a Prognosis About Recovery of Pain, Function, and Quality of Life After Rotator Cuff Repair: An Exploratory Longitudinal Study. J Orthop Sports Phys Ther. 2024 Aug;54(8):530-540. doi: 10.2519/jospt.2024.12398. PMID 39096935
- [Derived] Schwank A, Struyf T, Struyf F, Blazey P, Mertens M, Gisi D, Pisan M, Meeus M. Are psychosocial variables, sleep characteristics or central pain processing prognostic factors for outcome following rotator cuff repair? A protocol for a prospective longitudinal cohort study. BMJ Open. 2022 Aug 4;12(8):e058803. doi: 10.1136/bmjopen-2021-058803. PMID 35926993